CLINICAL TRIAL: NCT01478633
Title: Evaluation of Efficacy and Safety of Galantamine in Subjects With Dementia of Alzheimer's Type Who Failed to Benefit From Donepezil
Brief Title: Evaluation of Efficacy and Safety of Galantamine in Patients With Dementia of Alzheimer's Type Who Failed to Benefit From Donepezil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018649; JNS023-JPN-02 (Other: Janssen Pharmaceutical K. K., Japan)
Record Dates: First submitted 2011-11-03; First posted 2011-11-23 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Dementia; Galantamine; Donepezil
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galantamine (Experimental)
  Interventions: Drug: Galantamine

INTERVENTIONS:
Drug: Galantamine — 8 mg/day (4 mg twice daily) for 4 weeks, followed by 16 mg/day (8 mg twice daily) for an additional 4 weeks, followed by dose at 16 mg or increased to 24 mg (with the option of decreasing back to 16 mg) for the remainder of the study (to week 24)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of galantamine in patients who failed to benefit from donepezil (patients switching from donepezil). In clinical practice, it is expected that galantamine will be used in patients switching from donepezil due to the insufficient efficacy of donepezil.

DETAILED DESCRIPTION:
This is a nonrandomized (study drug is intentionally assigned), open-label (all people involved know the identity of the intervention), single-arm (one group of patients receiving the same treatment), multi-centered study of galantamine in patients with Alzheimer's disease (AD). Galantamine has been approved for treatment of mild to moderate dementia of AD. Galantamine is available as film-coated tablet in 68 countries including the United States and Europe, and is also available as oral syrup and extended-release capsule in 65 counties. In Japan, galantamine was approved in January 2011 and is available in three dosage forms of film-coated tablet, oral disintegrant tablet, and oral syrup. The target population is patients with mild to moderate dementia of Alzheimer's type (ie, Mini-Mental State Examination [MMSE] ranging from 10 to 22) who failed to benefit from donepezil. Patients must have diagnosis of probable AD according to the diagnostic criteria National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) study group. To ensure that at least 100 subjects complete the study, 125 subjects will be enrolled. The treatment group is to receive flexible dosing of 16 mg/day or 24 mg/day. Patients will receive the study treatment for 24 weeks in accordance with the dosing regimen specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of probable Alzheimer's disease (AD) in accordance with the diagnostic criteria of NINCDS-ADRDA study group
* Have an MMSE score of 10 to 22 inclusive at screening
* Have taken donepezil stably at 5 mg/day for more than 6 months before screening
* Have progression (worsening) of impaired cognitive function 6 months or longer before screening
* Be considered medically stable by the investigator on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Be medically stable on the basis of clinical laboratory tests performed at screening

Exclusion Criteria:

* Has any concurrent neurodegenerative diseases manifesting dementia other than Dementia of Alzheimer's type
* Has suspected impaired cognitive function due to a variety of causes
* Has significant health disorders or diseases according to the investigators' detailed criteria
* Has had major surgery within 52 weeks of screening, or will not have fully recovered from surgery, or planned surgery during the time the subject is expected to participate in the study
* Is a woman who is pregnant, or breast-feeding, or planning to become pregnant or is a man who plans to father a child while enrolled in this study
* Has a history of severe drug allergy or severe drug hypersensitivity
* Has a history of drug or alcohol abuse
* Used another investigational drug within 90 days of screening
* Used anti-dementia drugs marketed or being developed other than donepezil or medications containing the same active ingredients within 6 months of screening
* Is considered as ineligible by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The Change from Baseline in Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) Score at Week 24 | at Week 24
  The ADAS-J cog scale assesses memory, language and behavior and is composed of 11 tasks: word recall, spoken language ability, auditory comprehension, word finding difficulty in spontaneous speech, following commands, object and finger naming, constructional praxis, ideational praxis, orientation, word recognition, and recalling test instructions. The perfect total score is 70 points, and as the score becomes higher, the degree of impairment becomes severer.

SECONDARY OUTCOMES:
The Clinical Global Impression of Change (CGI-C) at Week 24 | at Week 24
  CGI-C is employed to evaluate the patient's global clinical improvement according to the rater's impression from 1 (Very much improved) to 7 (Very much worse).
Proportion of Responders at Week 24 | at Week 24
  Proportion of responders whose ADAS-J cog score at endpoint decreased from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K. K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (11):
- Japan (11):
  - Akita
  - Izunokuni
  - Kochi
  - Kumamoto
  - Osaka
  - Saitama
  - Takatsuki
  - Tokyo
  - Uji
  - Urayasu
  - Yokohama

REFERENCES:
- See also: Evaluation of Efficacy and Safety of Galantamine in Patients With Dementia of Alzheimer's Type Who Failed to Benefit From Donepezil — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3298&filename=JNS023-JPN-02_CSR.pdf